CLINICAL TRIAL: NCT02517307
Title: Role of Fatty Acid Oxidation Defects in Insulin Sensitivity
Brief Title: Fatty Acid Oxidation Defects and Insulin Sensitivity
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Oregon Health and Science University (Other)
Responsible Party: Principal Investigator, Melanie B Gillingham, Associate Professor, Oregon Health and Science University
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: OHSU11258
Record Dates: First submitted 2015-07-02; First posted 2015-08-07 (Estimated); Results first posted 2024-01-30 (Actual); Last update posted 2024-01-30 (Actual); Status verified 2023-12

CONDITIONS: Very Long-chain Acyl-CoA Dehydrogenase Deficiency; Trifunctional Protein Deficiency; Long-chain 3-hydroxyacyl-CoA Dehydrogenase Deficiency; Medium-chain Acyl-CoA Dehydrogenase Deficiency; Normal Volunteers; Carnitine Palmitoyltransferase II Deficiency, Myopathic
MeSH Terms: conditions — VLCAD deficiency; Trifunctional Protein Deficiency With Myopathy And Neuropathy; Medium chain acyl CoA dehydrogenase deficiency; Carnitine Palmitoyltransferase II Deficiency, Late-Onset | interventions — soybean oil, phospholipid emulsion; Heparin; Glycerol; Sodium Chloride

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- glycerol/saline FAOD (Experimental): Glycerol/Saline co-infusion hyperinsulinemic euglycemic clamp among subjects with a fatty acid oxidation disorder (FAOD)
  Interventions: Drug: Glycerol/Saline; Drug: Hyperinsulinemic euglycemic clamp
- intralipid FAOD (Experimental): Intralipid/Heparin co-infusion hyperinsulinemic euglycemic clamp among subjects with a fatty acid oxidation disorder (FAOD)
  Interventions: Drug: Intralipid/Heparin; Drug: Hyperinsulinemic euglycemic clamp
- glycerol/saline Control (Experimental): Glycerol/Saline co-infusion hyperinsulinemic euglycemic clamp among normal matched control subjects (control)
  Interventions: Drug: Glycerol/Saline; Drug: Hyperinsulinemic euglycemic clamp
- intralipid Control (Experimental): Intralipid/Heparin co-infusion hyperinsulinemic euglycemic clamp among normal matched control subjects (control)
  Interventions: Drug: Intralipid/Heparin; Drug: Hyperinsulinemic euglycemic clamp

INTERVENTIONS:
Drug: Intralipid/Heparin — Co-infusion of intralipid and heparin solutions during a hyperinsulinemic euglycemic clamp
  Arms: intralipid Control; intralipid FAOD
Drug: Glycerol/Saline — Co-infusion of a glycerol/saline solutions during a hyperinsulinemic euglycemic clamp
  Arms: glycerol/saline Control; glycerol/saline FAOD
Drug: Hyperinsulinemic euglycemic clamp — Infusion of insulin at at 40 mU/m2/min for 5 hours. Blood glucose will be monitored every 5 min during the insulin infusion and euglycemia will be maintained throughout the clamp by infusing 20% dextrose at a variable rate.

SUMMARY:
The purpose of this study is to learn more about what causes insulin resistance. It has been suggested that proper breakdown of fat into energy (oxidation) in the body is important to allow insulin to keep blood sugar in the normal range. The investigators want to know if having one of the fatty acid oxidation disorders could have an influence on insulin action. Fatty acid oxidation disorders are genetic disorders that inhibit one of the enzymes that converts fat into energy. The investigators will study both normal healthy people and people with a long-chain fatty acid oxidation disorder.

DETAILED DESCRIPTION:
The overall goal of this proposal is to investigate the effects of disordered mitochondrial fatty acid oxidation on insulin resistance in humans. Mitochondrial dysfunction has been implicated in the development of insulin resistance and type 2 diabetes during excess dietary fat intake and from increased release of endogenous free fatty acids , such as occurs in obesity. Controversy exists, however, as to whether this insulin resistance results from intrinsic defects in mitochondrial energy utilization or from abnormalities resulting from excess free fatty acid flux, as well as the role that subsequent accumulation of cellular metabolic intermediates play in impaired insulin signaling.

To address these controversies, the investigators will study a unique population of patients with inherited defects in each of the three mitochondrial enzymes in the fatty acid oxidation pathway: 1) very long-chain acyl-CoA dehydrogenase (VLCAD); 2) trifunctional protein (TFP, which includes long-chain 3-hydroxyacyl-CoA dehydrogenase (LCHAD)); and 3) medium-chain acyl-CoA dehydrogenase (MCAD). These proteins are required for the oxidation of sequentially shorter fatty acids . The investigators will test the hypothesis that intrinsic defects in mitochondrial function involving oxidation of long-chain, but not medium-chain, fatty acids are sufficient to prevent intralipid-induced insulin resistance.

ELIGIBILITY:
Inclusion Criteria:

* confirmed diagnosis of VLCAD, LCHAD, TFP or MCAD deficiency or same gender, age and BMI as a subject with a fatty acid oxidation disorder
* ability to travel to Oregon Health & Science University, Portland, Oregon
* ability and willingness to complete the protocol

Exclusion Criteria:

* hemoglobin <10g/dl, international normalized ratio (INR) >1.2 Prothrombin time (PTT) >36 sec, Platelets <150K/mm3
* pregnant or lactating females
* endocrine disorder such as diabetes or untreated thyroid disease
* cardiovascular disease or elevated plasma lipids
* regularly taking meds that strongly affect bleeding, bruising or platelets

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 41 (Actual)
Dates: Start 2016-02; Primary Completion 2021-01 (Actual); Study Completion 2021-03 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Oregon Health & Science University, Portland, Oregon, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 2 control participants were recruited between February 2016 and June 2016 to complete testing of the protocol procedures. Adjustments to clamp, MRS and biopsy protocols were made and a final manual of operating procedures developed. These 2 participants were not included in the final data analysis. Then, 23 participants with a FAOD were screened for eligibility from June 2016 to August 2019. 27 control participants were screened for eligibility from July 2016 to February 2020.
Pre-assignment Details: 2 initial control participants who did not have a comparable FAO matched participant completed the protocol procedures to establish the final protocol; the data was not included in the final analysis. 23 participants with a FAOD were randomized. Of those randomized, 2 did not meet inclusion criteria, and 2 declined to participate. 27 control participants were randomized. Of those randomized, 2 did not meet inclusion criteria and 3 declined to participate.
Groups:
- FAOD Glycerol Then Intralipid: Participants with a FAOD first complete a hyperinsulinemic euglycemic clamp with a co-infusion of glycerol. After a wash-out of 4 months, they then complete a a hyperinsulinemic euglycemic clamp with a co-infusion of intralipid.
- FAOD Intralipid Then Glycerol: Participants with a FAOD first complete a hyperinsulinemic euglycemic clamp with a co-infusion of intralipid. After a wash-out of 4 months, they then complete a a hyperinsulinemic euglycemic clamp with a co-infusion of glycerol.
- Control Glycerol Then Intralipid: Matched normal control participants first complete a hyperinsulinemic euglycemic clamp with a co-infusion of glycerol. After a wash-out of 4 months, they then complete a a hyperinsulinemic euglycemic clamp with a co-infusion of intralipid.
- Control Intralipid Then Glycerol: Matched normal control participants first complete a hyperinsulinemic euglycemic clamp with a co-infusion of intralipid. After a wash-out of 4 months, they then complete a a hyperinsulinemic euglycemic clamp with a co-infusion of glycerol.
Period: Overall Study
Arm/Group | FAOD Glycerol Then Intralipid | FAOD Intralipid Then Glycerol | Control Glycerol Then Intralipid | Control Intralipid Then Glycerol
Started | 11 | 8 | 11 | 11
Completed | 10 | 8 | 9 | 10
Not Completed | 1 | 0 | 2 | 1
Not completed — Withdrawal by Subject | 1 | 0 | 1 | 0
Not completed — Protocol Violation | 0 | 0 | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Control Glycerol Then Intralipid: Matched control participants first complete a hyperinsulinemic euglycemic clamp with a co-infusion of glycerol. After a wash-out of 4 months, they then complete a a hyperinsulinemic euglycemic clamp with a co-infusion of intralipid.
- Control Intralipid Then Glycerol: Matched control participants first complete a hyperinsulinemic euglycemic clamp with a co-infusion of intralipid. After a wash-out of 4 months, they then complete a a hyperinsulinemic euglycemic clamp with a co-infusion of glycerol.
- Total: Total of all reporting groups
Arm/Group | FAOD Glycerol Then Intralipid | FAOD Intralipid Then Glycerol | Control Glycerol Then Intralipid | Control Intralipid Then Glycerol | Total
Number analyzed (Participants) | 11 | 8 | 11 | 11 | 41
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 11 | 8 | 11 | 11 | 41
  >=65 years | 0 | 0 | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 32.0 (12.7) | 23.0 (4.3) | 33.8 (9.4) | 29.9 (10.8) | 29.32 (9.48)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 3 | 3 | 6 | 16
  Male | 7 | 5 | 8 | 5 | 25
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0 | 0
  Not Hispanic or Latino | 6 | 5 | 11 | 10 | 32
  Unknown or Not Reported | 5 | 3 | 0 | 1 | 9
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 1 | 1
  Asian | 0 | 0 | 0 | 1 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0 | 0
  White | 7 | 5 | 10 | 6 | 28
  More than one race | 0 | 0 | 0 | 1 | 1
  Unknown or Not Reported | 4 | 3 | 1 | 2 | 10
Region of Enrollment [Number; unit: participants]
  United States | 11 | 8 | 11 | 11 | 41

OUTCOME MEASURES:

1. Primary Outcome: Glucose Disposal Rate (Rd)- the Rate of Glucose Infusion to Maintain Euglycemia During Steady State Insulin Infusion in mg/Min
Description: Insulin infusion induces glucose disposal into muscle and adipose tissue in insulin sensitive participants. During the glycerol co-infusion, glucose disposal will be high. Intralipid co-infusion can induce a temporary insulin resistant state. During the intralipid co-infusion, glucose disposal will be decreased. We are comparing how intralipid dampens glucose disposal between participants with a FAOD and matched control participants. Glucose disposal is measured by measuring the ratio of deuterated glucose to unlabeled glucose at the beginning and end of the clamp. The calculated glucose disposal rate or RD is mg of glucose taken into muscle and adipose tissue per minute.
Time Frame: Calculated during the last 30 minutes of a 300 minute clamp.
Population: 1 participant with a FAOD withdrew after completing the glycerol clamp . 2 control participants completed the protocol to establish the study procedures, but are not included in the statistical analysis. 1 control participants withdrew and 1 was discontinued leaving 18 participants data for the intralipid clamp. In addition, 1 other control was discontinued and 1 control had technical challenges during the glycerol clamp leaving 16 control participants data for glycerol clamp.
Measure: Mean (Standard Deviation); unit: mg/min
Arm/Group | Glycerol/Saline FAOD | Intralipid FAOD | Glycerol/Saline Control | Intralipid Control
Number analyzed (Participants) | 19 | 18 | 16 | 18
mg/min | 709 (244) | 429 (297) | 842 (282) | 497 (297)
Statistical Analysis 1: Comparison: Glycerol/Saline FAOD vs Intralipid FAOD vs Glycerol/Saline Control vs Intralipid Control; We compared the effects of intralipid on Rd in controls subjects versus subjects with a FAOD by mixed-effect models. Factors were group (control or FAOD) treatment (glycerol or intralipid) and the interaction of those factors. The hypothesis was intralipid would decrease Rd in controls but not in subjects with an FAOD; Test type: Other; p = 0.136, Mixed Models Analysis

2. Secondary Outcome: Endogenous Glucose Production (Ra) - Calculated by the Equations of Steele During Steady State in mg/Min
Description: Infusion of insulin will suppress endogenous glucose production from the liver in insulin sensitive people. Insulin infusion with glycerol should suppress the endogenous glucose production in the liver but intralipid induces a temporary state of insulin resistance and the decrease in endogenous glucose production or Ra will be blunted with intralipid co-infusion. We are looking at the difference in Ra with intralipid between participants with a FAOD and matched control participants. Ra or endogenous glucose production during high insulin is measured in mg new glucose synthesized per minute.
Time Frame: Calculated during the last 30 minutes of a 300 minute clamp.
Population: 1 participant with a FAOD withdrew after completing the glycerol clamp . 2 control participants completed the protocol to establish the study procedures, but are not included in the statistical analysis. 1 control withdrew and 1 was discontinued leaving 18 participants data for the intralipid clamp. In addition, 1 other control was discontinued and 1 control had technical challenges during the glycerol clamp leaving 16 control participants data for the glycerol clamp.
Measure: Mean (Standard Deviation); unit: mg/min
Arm/Group | Glycerol/Saline FAOD | Intralipid FAOD | Glycerol/Saline Control | Intralipid Control
Number analyzed (Participants) | 19 | 18 | 16 | 18
mg/min | 84.7 (38.4) | 97.2 (44.0) | 50.2 (42.0) | 106 (37.0)
Statistical Analysis 1: Comparison: Glycerol/Saline FAOD vs Intralipid FAOD vs Glycerol/Saline Control vs Intralipid Control; We tested if intralipid did not suppress endogenous glucose production or Ra as much as glycerol in controls compared to subjects with an FAOD; Test type: Other — We analyzed the data with a mixed model looking at the effect of group (control vs FAOD) and treatment (glycerol vs intralipid) and their interaction; p = 0.011, Mixed Models Analysis

ADVERSE EVENTS:
Time Frame: 3 months for each intervention
Arm/Group | Glycerol/Saline FAOD | Intralipid FAOD | Glycerol/Saline Control | Intralipid Control
All-Cause Mortality (participants affected / at risk) | 0/19 | 0/18 | 0/20 | 0/21
Serious Adverse Events (participants affected / at risk) | 1/19 | 2/18 | 0/20 | 1/21
Other Adverse Events (participants affected / at risk) | 13/19 | 12/18 | 11/20 | 13/21
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Glycerol/Saline FAOD (N=19) | Intralipid FAOD (N=18) | Glycerol/Saline Control (N=20) | Intralipid Control (N=21)
Rhabdomyolysis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Urinary Tract Infection/Kidney Infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Glycerol/Saline FAOD (N=19) | Intralipid FAOD (N=18) | Glycerol/Saline Control (N=20) | Intralipid Control (N=21)
Headache (General disorders) | 3 (4) | 2 (2) | 1 (1) | 2 (2)
Pain at muscle biopsy site (Surgical and medical procedures) | 9 (9) | 9 (9) | 5 (5) | 5 (5)
Pain at fat biopsy site (Surgical and medical procedures) | 2 (2) | 1 (1) | 4 (4) | 2 (2)
Upper respiratory infection/colds (Infections and infestations) | 4 (4) | 2 (2) | 1 (1) | 2 (2)
UTI (Infections and infestations) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
allergic reaction (General disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Emesis, Diarrhea, GI upset, Nausea (Gastrointestinal disorders) | 1 (1) | 3 (3) | 3 (3) | 4 (5)
Hematoma at fat biopsy site (Surgical and medical procedures) | 2 (2) | 2 (2) | 3 (3) | 2 (2)
Bleeding or bruising at biopsy sites (Surgical and medical procedures) | 0 | 0 | 0 | 4 (6)
Tooth pain (General disorders) | 2 (2) | 0 | 0 | 0
Syncopal episode (Nervous system disorders) | 0 | 2 (2) | 0 | 0
general pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 3 (3) | 0 | 0
hypoglycemia during clamp (Endocrine disorders) | 0 | 0 | 1 (1) | 0
IV infiltration or phlebitis (Surgical and medical procedures) | 1 (1) | 0 | 1 (1) | 0
heavy menstrual cycles (Reproductive system and breast disorders) | 0 | 0 | 0 | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-03-23): https://cdn.clinicaltrials.gov/large-docs/07/NCT02517307/Prot_SAP_000.pdf